CLINICAL TRIAL: NCT06313372
Title: Interpreting Respiratory Oscillometry in Adult Asthma and COPD: a Delphi Study
Status: Not yet recruiting | Type: Observational
Sponsor: Scius Healthcare Solutions Pty Ltd (Industry)
Collaborators: Chiesi Australia (Unknown)
Responsible Party: Sponsor
Other Study IDs: CA2085
Record Dates: First submitted 2024-02-26; First posted 2024-03-15 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
Keywords: Respiratory oscillometry; Impulse oscillometry; Forced oscillation technique
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Respiratory oscillometry — This a Delphi study where we are obtaining expert opinion and input on the use of respiratory oscillometry (a diagnostic respiratory test) in the assessment and management of patients with asthma or chronic obstructive pulmonary disease. The participants are respiratory specialists/pulmonologists. They are sharing their insights into the clinical use of respiratory oscillometry via a series of online surveys. The Delphi process is used in an attempt to achieve consensus as to how respiratory oscillometry is used in clinical practice. As such there is no intervention being used on the study participants, but they are sharing insights on how the respiratory test is used in their clinical practice in order to obtain consensus on this use.

SUMMARY:
This is an international Delphi study to consolidate expert consensus on the use of respiratory oscillometry in the management of adult patients with asthma or chronic obstructive pulmonary disease (COPD).

The primary objective of the Delphi study is to aid the interpretation of respiratory oscillometry in clinical practice amongst adult patients with asthma or COPD. This will be achieved by obtaining expert consensus on:

* Which parameters are used in clinical practice for impulse oscillometry (IOS) and for forced oscillation technique (FOT) devices.
* What cut-offs can be used for each parameter to guide clinical practice in the management of adult patients with asthma and COPD.

This study is based on the Delphi methodology. The Delphi study will comprise of four rounds, one brainstorming round, to formulate the consensus survey, and three rounds to attempt to obtain consensus.

In each round a questionnaire comprising of statements and questions regarding respiratory oscillometry will be sent to participants in the Delphi study electronically using SurveyLet, an online survey platform. Participants will respond anonymously to the survey questions, indicating their level of agreement or disagreement with each statement or question. Participants will be given 4 weeks to complete each round of the Delphi study.

Questions and statements will be repeated in subsequent rounds until the predefined level of consensus is met or the maximum number of rounds is achieved (limited to a maximum of 3 rounds). Aggregated results for each statement or question, including distribution of results and consensus status, will be provided to participants after each round to facilitate informed decisions in subsequent rounds.

DETAILED DESCRIPTION:
Study procedures:

The Delphi study will comprise of four rounds, one brainstorming round and three rounds to attempt to obtain consensus.

A series of anonymous questionnaires will be administered to a panel of experts and respiratory specialists familiar with oscillometry testing.

Phase one: Brainstorming to develop survey questionnaire.

The initial brainstorming questionnaire will be developed by the Steering Committee, based on the published literature and clinical practice. The brainstorming questionnaire will be circulated to a selected group of respiratory specialists who are known experts in respiratory oscillometry for refinement and testing.

The expert panel will comprise of approximately 10 respiratory specialists who have published papers on respiratory oscillometry. This brainstorming questionnaire will be open in nature and will allow all respondents to propose new statements as well as adjust the proposed statements that are to be evaluated by their peers.

The results of the brainstorming round will be reviewed by the Steering Committee to finalise the questionnaire for the first round of the Delphi study.

Phase two: Attempting to achieve consensus.

To obtain consensus three iterative rounds (Rounds 1-3) will be undertaken. In each round a questionnaire comprising of statements and questions regarding respiratory oscillometry will be sent to all participants in the Delphi study electronically using SurveyLet, an online survey platform utilising the Delphi technique.

The initial questionnaire for use in Round 1, will be the survey developed in the brainstorming round.

There will be a range of statement types used to ascertain consensus, including:

* Agreement with statements ranked using a six-point scale (Agree Strongly', ''Agree Moderately', Agree Slightly', 'Disagree Slightly', 'Disagree Strongly', ''Disagree Moderately').
* Agreement on importance/clinical utility of various oscillometry parameters using a ranking process.
* Agreement on defining values (cut-offs) for clinically relevant changes for the various oscillometry parameters.

Participants will be encouraged to provide free text comments after each statement or question and these comments will be reviewed by the Steering Committee to determine if the questionnaire needs revision prior to the next survey round.

Questions and statements will be repeated in subsequent rounds until the predefined level of consensus is met or the maximum number of rounds is achieved (limited to a maximum of 3 rounds).

Aggregated results for each statement or question, including distribution of results and consensus status, will be provided to participants after each round to facilitate informed decisions in subsequent rounds.

Participants will be given 4 weeks to complete each round of the Delphi study. During a Delphi study, participants with a minority opinion can become discouraged and drop out of the study, potentially resulting in an overestimation of consensus.

At the commencement of the study, participants will be sent an email with an encrypted personalised secure link (to the study questionnaire). This secure link means that each participant can only view their own data and the aggregated data shared in study rounds 2 and 3. No study participant nor the lead investigators can see the individual responses of any other participant. Access to subsequent study rounds is also via the encrypted secure link or via the participant login into the SurveyLet platform.

In this study, consensus is achieved when ≥ 70% of the participants give the same answer for any question or statement.

For questions and statements that are assessed using a 6-point agreement scale, consensus is achieved when ≥ 70% of participants either:

* 'Agree Strongly' or ''Agree Moderately'
* 'Agree Slightly' or ''Disagree Slightly'
* 'Disagree Strongly' or ''Disagree Moderately'

For questions and statements that are assessed using a ranking process, consensus is achieved when ≥ 70% of participants give that ranking.

For questions and statements that are assessed using a defined value, consensus is achieved when ≥ 70% of participants give the same value.

ELIGIBILITY:
Inclusion Criteria:

* Respiratory specialist in active clinical practice ≥ 12 months.
* Use respiratory oscillometry ≥ 2 tests per week

Exclusion Criteria:

* Only use respiratory oscillometry when participating in clinical trials
* Employee or stockholder of pharmaceutical company
* Employee or stockholder of oscillometry manufacturer
* Employee or stockholder of tobacco/vaping companies.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants in the Delphi study will be respiratory specialists with expertise in the application of respiratory oscillometry in clinical practice and who routinely use respiratory oscillometry in clinical practice. Clinical use is defined as respiratory specialists who order and/or interpret respiratory oscillometry in day-to-day clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Identification of which respiratory oscillometry parameters (resistance, [R5, R20, R5-R20], reactance [X5, delta X5] or reactance area [AX]) are used to guide clinical management of asthma or COPD as determined by expert consensus using a ranking scale. | When consensus is achieved within an individual Delphi round or through to study end, up to 1 year
  Participants are asked to rank in order of clinical importance the different respiratory oscillometry parameters (R5, R20, X5, AX, R5-R20, delta X5) from 1 to 6
  Consensus is achieved when ≥ 70% of the participants give the same ranking order within an individual round of the Delphi study. If consensus is not achieved, aggregated data from the previous round is shared and the participants are asked to provide their ranking again.
Identification of cut-off values used for respiratory oscillometry parameters (R5, X5, AX, R5-R20) to define an abnormal test result as determined by expert consensus using a 6-point categorical scale (Agree strongly to Disagree strongly) | When consensus is achieved within an individual Delphi round or through to study end, up to 1 year
  Cut-off values used to define abnormality are proposed for each parameter (R5, X5, AX, and R5-R20) and the participants/experts are asked for their level of agreement with the proposed cut-off value being assessed.
  An example of the type of statement used for this component of the survey is as follows:
  For R5, a result with a z-score > 1.64 is considered abnormal.
  A. Agree Strongly B. Agree Moderately C. Agree Slightly D. Disagree Slightly E. Disagree Moderately F. Disagree Strongly
  Consensus is achieved when ≥ 70% of the participants give the same level of agreement for each statement within an individual round of the Delphi study. If consensus is not achieved, aggregated data from the previous round is shared and the participants are asked to provide their level of agreement again.

SECONDARY OUTCOMES:
Identification of cut-off values used for respiratory oscillometry parameters (R5, X5, and AX) to define a bronchodilator response as determined by expert consensus using a 6-point categorical scale (Agree strongly to Disagree strongly) | When consensus is achieved within an individual Delphi round or through to study end, up to 1 year
  Cut-off values used to define a bronchodilator response are proposed for each parameter (R5, X5, and AX) and the participants/experts are asked for their level of agreement with the proposed cut-off value being assessed.
  An example of the type of statement used for this component of the survey is:
  For R5, a result with a z-score > 1.4 is considered to be a significant bronchodilator response.
  A. Agree Strongly B. Agree Moderately C. Agree Slightly D. Disagree Slightly E. Disagree Moderately F. Disagree Strongly
  Consensus is achieved when ≥ 70% of the participants give the same level of agreement for each statement within an individual round of the Delphi study. If consensus is not achieved, aggregated data from the previous round is shared and the participants are asked to provide their level of agreement again.
Identification of cut-off values used for oscillometry parameters (R5, X5, AX, R5-R20) to define a significant clinical change between visits as determined by expert consensus using a 6-point categorical scale (Agree strongly to Disagree strongly) | When consensus is achieved within an individual Delphi round or through to study end, up to 1 year
  Cut-off values used to define a significant clinical change between visits are proposed for each parameter (R5, X5, AX and R5-R20) and the participants/experts are asked for their level of agreement with the proposed cut-off value being assessed.
  An example of the type of statement used for this component of the survey is:
  For R5, a result with a z-score > 0.5 is considered a significant change between visits.
  A. Agree Strongly B. Agree Moderately C. Agree Slightly D. Disagree Slightly E. Disagree Moderately F. Disagree Strongly
  Consensus is achieved when ≥ 70% of the participants give the same level of agreement for each statement within an individual round of the Delphi study. If consensus is not achieved, aggregated data from the previous round is shared and the participants are asked to provide their level of agreement again.

CONTACTS AND LOCATIONS:
Overall Officials: Li Ping Chung, MBBS, Principal Investigator — Fiona Stanley Hospital

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other study participants as a fundamental aspect of a Delphi study is that any data shared during the Delphi process is anonymous and therefore professional reputation does not introduce bias into the achievement of consensus.
  Anonymized (excluding individual demographics that jeopardise participant privacy) aggregated data will be shared on an appropriate public platform at the time of publication.